CLINICAL TRIAL: NCT07352111
Title: High-risk Coronary Atherosclerosis in Subjects With Family History of Myocardial Infarction; the FAMILY Study
Brief Title: High-risk Coronary Atherosclerosis in Subjects With Family History of Myocardial Infarction
Acronym: FAMILY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Principal Investigator, Elena Cittera, Director, I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FAMILY Study
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Diease
Keywords: Cardiac CT; family history of CAD; atherosclerosis; primary prevention
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac CT in primary prevention (Experimental): Patients asymptomatic but with family history of CAD will undergo cardiac CT with advance plaque evaluation
  Interventions: Diagnostic Test: Cardiac CT

INTERVENTIONS:
Diagnostic Test: Cardiac CT — Cardiac CT with advance plaque evaluation will be performed

SUMMARY:
The evidence of high-risk atherosclerosis at cardiac CT (CCT) may support aggressive primary prevention treatment, reducing the risk of future cardiovascular events. Family history of coronary artery disease (CAD) is a risk factor for cardiovascular events but limited data described the prevalence of coronary atherosclerosis in these patients.

Aims of the FAMILY project are to explore the prevalence of high-risk coronary atherosclerosis among patients with family history of CAD, to explore whether CCT in this setting may to reclassify patients' vs standard of care and to explore correlations between genetic background and high risk and potentially unstable coronary atherosclerosis.

A consecutive cohort of asymptomatic of patients with family history of CAD will be prospectively enrolled. A per-protocol CCT with advanced atherosclerosis analysis will be performed. At the time of CCT a blood sample will be collected for bio-humoral and genetic investigation. The prevalence of high risk atherosclerosis will be quantified, the reclassification rate of CCT vs clinical evaluation evaluated and the potential in vivo association between genetic profile and high risk atherosclerosis explored.

ELIGIBILITY:
Inclusion Criteria:

* patients with postive family history of CAD

Exclusion Criteria:

* known cardiovascular diseases
* any symptoms

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk reclassification | 3 years
  Risk reclassification rate will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Galeazzi-Sant'Ambrogio IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No